CLINICAL TRIAL: NCT02119234
Title: Open-label, Randomized, 3-way Cross-over, Placebo Controlled, Single Dose Clinical Pharmacology Study in COPD Patients After Inhalation of CHF 5993 pMDI Using the Standard Actuator With or Without AeroChamber Plus Flow-Vu VHC Spacer
Brief Title: Pharmacokinetics of CHF 5993 pMDI With and Without Spacer in COPD Patients
Acronym: TRIPLE 4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-05993AA1-04; 2013-003770-27 (EudraCT Number)
Record Dates: First submitted 2014-04-11; First posted 2014-04-21 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Beclomethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CHF5993 pMDI + Spacer (Experimental): CHF 5993 pMDI (Beclometasone/formoterol/glycopyrrolate 100/6/25 mcg per actuation) x 4 inhalations administered using Aerochamber Plus Flow-vu VHC spacer
  Interventions: Drug: Beclometasone/formoterol/glycopyrrolate
- CHF5993 pMDI (Active Comparator): CHF 5993 pMDI (Beclometasone/formoterol/glycopyrrolate 100/6/25 mcg per actuation) x 4 inhalations administered using standard actuator only
  Interventions: Drug: Beclometasone/formoterol/glycopyrrolate
- Placebo pMDI (Placebo Comparator): Placebo pMDI x 4 inhalations
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Beclometasone/formoterol/glycopyrrolate
  Other Names: CHF5993 pMDI
  Arms: CHF5993 pMDI; CHF5993 pMDI + Spacer
Drug: Placebo
  Arms: Placebo pMDI

SUMMARY:
The study is performed to investigate the effect of the spacing device on the pharmacokinetics of CHF 5993 pMDI active ingredients administered with and without Aerochamber Plus Flow-vu antistatic VHC spacer as a single administration in COPD patients. Moreover, the general safety and tolerability of the treatments will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients
* smokers or ex-smokers
* post-bronchodilator FEV1 between 30 and 60% of predicted value

Exclusion Criteria:

* Positive serology to HIV and hepatitis
* Known respiratory disorder other than COPD
* Recent COPD exacerbations or hospitalization for COPD
* Treatment with non-permitted concomitant medication
* clinically relevant concomitant disease
* clinically relevant abnormal laboratory or ECG parameters

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Area under the curve of B17MP, formoterol and glycopyrrolate | Over 24 and 48h after single administration
  AUCt (up to the last quantifiable concentration) and Cmax (maximum concentration) from plasma concentrations vs time profiles.
  over 24h for formoterol and B17MP, over 48h for glycopyrrolate

SECONDARY OUTCOMES:
Other pharmacokinetic parameters for formoterol, glycopyrrolate and B17MP in plasma | over 24 or 48h after single administration
  B17MP AUC0-30min, AUC0-24h, AUCinf, tmax, half-life Formoterol AUC0-30min, AUC0-24h, AUCinf, tmax, half-life Glycopyrrolate AUC0-30min, AUC0-48h, AUCinf, tmax, half-life
Adverse events | over a period of 6 to 11 weeks
  from the signature of the informed consent until the follow-up phone call
Lung function | 30 min after single administration
  FEV1
plasma cortisol | over 24 h after single administration
  cortisol AUC0-24h, Cmin and tmin
cortisol urinary excretion | over 24 h after single administration
  cortisol excretion corrected and not corrected for creatinine
potassium plasma profile | over 24 h after single administration
  potassium AUC0-24h, tmin and Cmin
Vital signs | over 24 h after single administration
  systolic and diastolic blood pressure
ECG parameters | over 24 h after single administration
  extracted from holter recording HR, QTcF, PR and QRS

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kuna, MD, Principal Investigator — Medical University Lodz
Locations (1):
- Medical University in Lodz, Lodz, Ul. Kopcińskiego 22, Poland

REFERENCES:
- See also: CSR Synopsis available in the Chiesi Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_CCD-05993AA1-04.pdf